CLINICAL TRIAL: NCT00715091
Title: Effects of NSAIDs on RAdiographic Damage in Ankylosing Spondylitis (ENRADAS) - a Prospective Randomised Controlled Trial
Brief Title: Effects of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) on RAdiographic Damage in Ankylosing Spondylitis
Acronym: ENRADAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, J. Sieper, Prof., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENRADAS-01; EUDA-CT: 2007-007637-39
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Ankylosing Spondylitis
Keywords: NSAIDS; ankylosing spondylitis; SpA; Spondyloarthritis; radiographic changes
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): continuous (daily) treatment with diclofenac cholestyramine 150 mg (Voltaren Resinate), divided into 75mg Voltaren twice daily
  Interventions: Drug: diclophenac
- 2 (Active Comparator): treatment on-demand (as needed) with diclofenac-cholestyramine 75 to 150 mg (Voltaren Resinate). The treatment strategy of the control intervention (on-demand) reflects current clinical practice in AS.
  Interventions: Drug: diclophenac

INTERVENTIONS:
Drug: diclophenac — continuous (daily) treatment of diclofenac cholestyramine 150 mg, divided into 75mg twice daily
  Other Names: voltaren resinat
  Arms: 1
Drug: diclophenac — treatment on-demand (as needed) with diclofenac-cholestyramine 75 to 150 mg daily
  Other Names: Voltaren resinate
  Arms: 2

SUMMARY:
This is a randomised, controlled, multi-centre clinical trial on AS patients. Experimental intervention: continuous (daily) treatment with diclofenac cholestyramine 150 mg (Voltaren Resinate), divided into 75mg Voltaren twice dailyControl intervention: treatment on-demand (as needed) with diclofenac-cholestyramine 75 to 150 mg (Voltaren Resinate). The treatment strategy of the control intervention (on-demand) reflects current clinical practice in AS. Duration of intervention per patient: 2 years Follow-up per patient: safety assessment 3 months after termination of the trial.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a common chronic inflammatory rheumatic disease with a prevalence of about 0.5%. First symptoms normally occur in young adulthood. Early in its course, AS is dominated by chronic pain, fatigue and morning stiffness, later on by ankylosis and loss of function. Nonsteroidal anti-inflammatory drugs (NSAID) and tumor necrosis factor (TNF) alpha blocking agents are the only drugs with proven efficacy for signs and symptoms. It is not clear, however, whether these drugs are also capable of retarding or stopping structural damage, i.e. prevention of bony ankylosis. Earlier investigations indicated that NSAIDs have, in addition to their anti-inflammatory, also an anti-osteoproliferative effect. In this study we will investigate whether treatment with 150 mg diclofenac, a non-selective NSAID, on a daily basis (continuous treatment) over 2 years is capable to slow down the development of bony ankylosis as compared to treatment with 75-150mg diclofenac as needed according to clinical symptoms (on-demand treatment). In this national multi-centre randomized trial patients with symptomatic AS and indication for NSAID therapy will be enrolled in about 40 centres. The primary outcome parameter is the proportion of patients with radiographic progression in the spine after 2 years in each treatment arm. If continuous NSAID treatment results in less radiographic progression as compared to on-demand treatment, a true disease modifying effect of NSAID has to be assumed which will most likely change the place of NSAID treatment in AS.

ELIGIBILITY:
Inclusion Criteria:

* AS according to mod. New York criteria
* Patients must have radiographic damage (at least one syndesmophyte) of the spine but no complete ankylosis of the cervical and lumbar spine (these are patients at risk for further and more rapid radiographic progression)
* Patients must have active disease at inclusion defined as BASDAI question 2 (related to back pain) >= 4 (VAS, range 0-10) without NSAID treatment and with a clinical indication for NSAID therapy based on signs and symptoms

Exclusion Criteria:

* No radiographic damage (syndesmophyte) of the spine at baseline
* Complete ankylosis of the cervical and lumbar spine
* Inactive disease
* Evidence of current or past peptic ulcer
* Current or past coronary heart disease
* Stroke or transient ischemic attack
* Uncontrolled hypertension
* Chronic renal failure (creatinine > 1.5mg/dl)
* Impaired liver function
* Pregnancy
* Abnormal liver function (2x upper limit of normal)
* Active hepatitis B or C, chronic or acute heart failure (NYHA III or IV) -
* History of HIV infection
* History of neoplastic disease (details please refer to exclusion criteria)
* History of abuse of "hard" drugs or alcoholism
* Concomitant treatment with steroids, TNF-blockers, other DMARDs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
radiographic change (mean) of the spine after 2 years in the per-protocol population. Radiographs will be collected and centrally digitized. Scoring will be done by 2 readers who were blinded to treatment and sequence of the films | 2 years

SECONDARY OUTCOMES:
the proportions of patients with any progression (change in the mSASSS ≥ 1) and change in the mSASSS > smallest detectable change (SDC), i.e. change in mSASSS which is greater than the measurement error. | 2 years
ITT analysis of radiographic change. | 2 years
Change in VAS back pain, BASDAI, BASFI, BASMI, CRP. | 2 years
event rates of serious and non-serious adverse events will be documented and compared between the two groups. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rudwaleit, MD, Principal Investigator — Charité University, Berlin, Germany; Joachim Sieper, MD, Principal Investigator — Charité University, Berlin, Germany; Jürgen Braun, MD, Principal Investigator — Rheumazentrum Ruhrgebiet, Herne, Germany
Locations (30):
- Germany (30):
  - Medizinische Universitätsklinik Innere Medizin, Tübingen, Baden-Wurttemberg
  - Praxis Dr. Jacki, Tübingen, Baden-Wurttemberg
  - Praxis Dr. Manger, Bamberg, Bavaria
  - Praxis Dr. Ochs, Bayreuth, Bavaria
  - Praxis Dr. Kellner, München, Bavaria
  - Praxiszentrum St. Bonifazius, München, Bavaria
  - Gemeinschaftspraxis Dr. Göttl, Passau, Bavaria
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Praxis Dr. Rockwitz, Goslar, Lower Saxony
  - Gemeinschaftspraxis Dr. von Hinüber, Hildesheim, Lower Saxony
  - Gemeinschaftspraxis Dr. Gauler, Osnabrück, Lower Saxony
  - Praxis Dr. Dockhorn, Weener, Lower Saxony
  - Universitätsklinikum DüsseldorfKlink für Endokrinologie, Diabetologie und Rheumatologie, Düsseldorf, North Rhine-Westphalia
  - Rheumatologische Schwerpunktpraxis, Düsseldorf, North Rhine-Westphalia
  - Evangelisches Krankenhaus, Ratingen, North Rhine-Westphalia
  - Praxis Dr. Kramer, Remscheid, North Rhine-Westphalia
  - Praxis Dr. Schoo, Rheine, North Rhine-Westphalia
  - Rheumatologische Praxis Dr. Spieler, Zerbst, Saxony-Anhalt
  - Brandt, Berlin
  - Praxis Mielke, Berlin
  - Praxis Zinke, Berlin
  - Gemeinschaftspraxis Dr. Schwenke, Dresden
  - Praxis Dr. Pick, Grafschaft Bei Bad Neuenahr-Ahrweiler
  - Praxis Dr. Kühne, Haldensleben I
  - Rheumazentrum Ruhrgebiet, St. Josefs Krankenhaus, Herne
  - St. Josefs-Krankenhaus, Rheumatologie, Herne
  - Praxis Dr. Kapelle, Hoyerswerda
  - Gemeinschaftspraxis Dr. Kolitsch, Katzhütte
  - Praxis Dr. Gräßler, Pirna
  - Praxis Bohl-Bühler, Potsdam

REFERENCES:
- [Background] Wanders A, Heijde Dv, Landewe R, Behier JM, Calin A, Olivieri I, Zeidler H, Dougados M. Nonsteroidal antiinflammatory drugs reduce radiographic progression in patients with ankylosing spondylitis: a randomized clinical trial. Arthritis Rheum. 2005 Jun;52(6):1756-65. doi: 10.1002/art.21054. PMID 15934081
- [Derived] Hartl A, Sieper J, Syrbe U, Listing J, Hermann KG, Rudwaleit M, Poddubnyy D. Serum levels of leptin and high molecular weight adiponectin are inversely associated with radiographic spinal progression in patients with ankylosing spondylitis: results from the ENRADAS trial. Arthritis Res Ther. 2017 Jun 15;19(1):140. doi: 10.1186/s13075-017-1350-9. PMID 28619118
- [Derived] Sieper J, Listing J, Poddubnyy D, Song IH, Hermann KG, Callhoff J, Syrbe U, Braun J, Rudwaleit M. Effect of continuous versus on-demand treatment of ankylosing spondylitis with diclofenac over 2 years on radiographic progression of the spine: results from a randomised multicentre trial (ENRADAS). Ann Rheum Dis. 2016 Aug;75(8):1438-43. doi: 10.1136/annrheumdis-2015-207897. Epub 2015 Aug 4. PMID 26242443